CLINICAL TRIAL: NCT03470701
Title: Improving Albuminuria Screening Compliance Using a Smartphone Urinalysis Kit in the Hypertensive Non-Diabetic Population
Brief Title: Improving Albuminuria Screening Compliance Using a Smartphone Urinalysis Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Kidney Foundation, United States (Other); Healthy.io Ltd. (Industry)
Responsible Party: Principal Investigator, Alexander Chang, Assistant Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2017-0516
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Albuminuria; Chronic Kidney Diseases; Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Albuminuria; Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - usual care (No Intervention): This arm will receive usual care.
- Mailed Urinalysis Smartphone Kit (Experimental): This arm will receive a mailed urinalysis smartphone kit if they do not complete albuminuria screening after the initial reminder to do so.
  Interventions: Other: Mailed Urinalysis Smartphone Kit

INTERVENTIONS:
Other: Mailed Urinalysis Smartphone Kit — Patients who fail to complete albuminuria screening after the initial reminder to do so, will be contacted by phone and offered a mailed smartphone urinalysis kit. Agreeable patients will then receive the mailed kit and instructions to use their smartphone camera to analyze a urine dipstick.
  Arms: Mailed Urinalysis Smartphone Kit

SUMMARY:
This study will test the effectiveness of mailed, smartphone urinalysis kits to improve albuminuria screening compliance and detection of albuminuria.

DETAILED DESCRIPTION:
This proposal will examine the effect of mailed, smartphone urinalysis kits to improve albuminuria screening compliance and detection of albuminuria. The investigators will randomize 1,000 non-diabetic MyGeisinger portal users with hypertension and last clinic blood pressure >= 130/80 mmHg who have not received albuminuria screening to either: 1) control - usual care or 2) intervention - mailed urinalysis smartphone kit. All patients will first receive a reminder letter to have albuminuria screening completed at their clinic in coordination with the Geisinger Care Gap Team. Patients randomized to the intervention arm who do not complete this initial screening test will then be offered a mailed, smartphone urinalysis testing kit. Patients with 1+ or greater detected urine protein will be recommended to have urine albumin/creatinine ratio (ACR) testing to confirm albuminuria. Patients with ACR >= 30 mg/g will be referred to pharmacists for optimal treatment of albuminuria (ACE or ARB, statin, BP goal <130/90 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Hypertension
* Last outpatient BP ≥ 130/80 mmHg
* Active MyGeisinger users with a listed mobile phone number
* Has a Geisinger PCP and followed by the Care Gaps team
* No prior urine albuminuria test (urine dipstick, albumin/creatinine ratio, protein/creatinine ratio)

Exclusion Criteria:

* History of diabetes
* Receiving dialysis
* History of kidney transplant
* eGFR < 15 ml/min/1.73m2
* Principal investigator or PCP discretion (i.e. concerns about safety, compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Completion of albuminuria screening | Baseline to 3 months of enrollment date
  Includes completion of mailed smartphone urinalysis and clinical labs (urinalysis, albumin/creatinine ratio, or protein/creatinine ratio)
Total number of detected albuminuria cases | Baseline to 3 months of enrollment date
  confirmed by urine albumin/creatinine ratio >= 30 mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Chang, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
May be available upon request

REFERENCES:
- [Derived] Leddy J, Green JA, Yule C, Molecavage J, Coresh J, Chang AR. Improving proteinuria screening with mailed smartphone urinalysis testing in previously unscreened patients with hypertension: a randomized controlled trial. BMC Nephrol. 2019 Apr 18;20(1):132. doi: 10.1186/s12882-019-1324-z. PMID 30999886